CLINICAL TRIAL: NCT06980584
Title: Analysis of Clinical Characteristics and Follow-Up Study on Treatment of Nonthrombotic Obstructive Pulmonary Hypertension: Interventional Study
Brief Title: Study on the Treatment of Nonthrombotic Obstructive Pulmonary Hypertension
Acronym: ACCT-NOPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KE-61_Int
Record Dates: First submitted 2025-04-27; First posted 2025-05-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-02

CONDITIONS: Fibrosing Mediastinitis; Pulmonary Hypertension
Keywords: Rituximab; Endobronchial Ultrasound; Pulmonary Vascular Intervention
MeSH Terms: conditions — Mediastinal Fibrosis; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combined treatment group (Experimental): Participants assigned to this group will receive both pulmonary vascular intervention and rituximab lymph node injection.
  Interventions: Procedure: Rituximab Lymph Node Injection Combined with Pulmonary Vascular Intervention
- Interventional-only group (Active Comparator): Participants assigned to this group will receive pulmonary vascular intervention alone.
  Interventions: Procedure: Pulmonary Vascular Interventional Therapy

INTERVENTIONS:
Procedure: Rituximab Lymph Node Injection Combined with Pulmonary Vascular Intervention — Based on the degree of vascular stenosis, individualized and periodic pulmonary vascular interventions are performed to reopen obstructed vessels. During the treatment cycle, one lymph node drug injection is administered: 50mg of rituximab is dissolved in 15ml of 5% glucose solution and injected at multiple sites into the identified enlarged mediastinal lymph nodes under ultrasound-guided bronchoscopy.
  Arms: Combined treatment group
Procedure: Pulmonary Vascular Interventional Therapy — According to the degree of vascular stenosis, individualized and periodic pulmonary vascular interventions are performed to reopen obstructed pulmonary vessels.
  Arms: Interventional-only group

SUMMARY:
Through a randomized controlled trial (RCT) design, this study aiming to evaluated the efficacy and safety of rituximab lymph node injection combined with pulmonary vascular interventional therapy in treating fibrosing mediastinal pulmonary hypertension (FM-PH).Eligible participants were randomly assigned to either the combined treatment group, receiving both pulmonary vascular intervention and rituximab lymph node injection, or the interventional-only group, which received pulmonary vascular intervention alone. At 3, 6, and 12 months post-treatment, the efficacy was assessed based on symptom improvement, hemodynamic changes, lesion volume reduction, etc. Safety was mainly evaluated by comparing adverse event incidence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with fibrosing mediastinitis between November 2024 and November 2026, aged between 18 and 85 years.
2. The patient presented with symptoms of chest tightness, shortness of breath, and reduced exercise tolerance.
3. Chest CT revealed mediastinal lymph node compression of the pulmonary artery, with evidence of pulmonary hypertension consistent with the patient's symptoms.
4. The subject signed the informed consent form prior to participation and is able to comply with the study protocol and one-year follow-up.

Exclusion Criteria:

1. Currently in the active phase of infection, including but not limited to tuberculosis, Histoplasma capsulatum, and Aspergillus infections;
2. The underlying primary disease, such as sarcoidosis, Behcet's disease, or uncontrolled IgG4-related disease, is currently not well controlled.
3. Before treatment, a large amount of pleural effusion was still present.
4. Pulmonary function tests (PFT) showed FEV1 <30% of the predicted value, FEV1/FVC <30%, and DLCO <30%.
5. There are contraindications to bronchoscopy or endovascular intervention.
6. Complicated by other end-stage organ dysfunction, such as Child-Pugh class C liver function or stage IV chronic renal failure.
7. Complicated by severe immunosuppression.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Six Minutes Walk Distance at 12 Months. | From enrollment to the end of treatment at 12 months
  Conduct 6-minute walk test to measure the 6-minute walk distance, and compare the walking distances at baseline and 12 months after treatment.
The incidence of treatment-related serious adverse events (SAE) | During the one-year follow-up period after treatment completion
  The incidence of treatment-related serious adverse events is measured by tracking and documenting any SAEs that occur during the treatment period, as well as through follow-up assessments. Each event is evaluated for severity and causality, and the incidence is calculated by dividing the number of patients who experience at least one treatment-related SAE by the total number of treated patients.

SECONDARY OUTCOMES:
Change from baseline in the World Health Organization Functional Classification of Pulmonary Hypertension at 3, 6 and 12 months. | From enrollment to the end of treatment at 3, 6 and 12 months.
  Change from Baseline in the World Health Organization Functional Classification of Pulmonary Hypertension (WHO-FC) which assessed based on clinical symptoms and signs at baseline and the end of treatment at 3, 6 and 12 months. The WHO-FC system consists of four levels: I, II, III, and IV. Higher levels indicate progressively more severe conditions.
Change from Baseline in the mean pulmonary artery pressure (mPAP) at 3 and 12 Months. | From enrollment to the end of treatment at 3 and12 months
  The mean pulmonary artery pressure (mPAP) was measured by right heart catheterization to evaluate the hemodynamic change from baseline to the end of treatment at 3 and12 months.
Change from Baseline in the Cardiac Index (CI) at 3 and 12 Months. | From enrollment to the end of treatment at 3 and12 months
  The Cardiac Index (CI) was measured by right heart catheterization to evaluate the hemodynamic change from baseline to the end of treatment at 3 and12 months.
Change from Baseline in the Pulmonary Vascular Resistance (PVR) at 3 and 12 Months. | From enrollment to the end of treatment at 3 and12 months
  The Pulmonary Vascular Resistance (PVR) was measured by right heart catheterization to evaluate the hemodynamic change from baseline to the end of treatment at 3 and12 months.
Change from Baseline in the forced vital capacity (FVC) at 3, 6 and 12 Months. | From enrollment to the end of treatment at 3, 6 and 12 months
  Pulmonary function tests was performed, including the forced vital capacity (FVC), to evaluated pulmonary function at baseline and the end of treatment at 3, 6 and 12 Months.
Change from Baseline in the forced vital capacity of predicted (FVC%pred) at 3, 6 and 12 Months. | From enrollment to the end of treatment at 3, 6 and 12 months
  Pulmonary function tests was performed, including the forced vital capacity of predicted (FVC%pred), to evaluated pulmonary function at baseline and the end of treatment at 3, 6 and 12 Months.
Change from Baseline in the forced expiratory volume in 1 second (FEV1) at 3, 6 and 12 Months. | From enrollment to the end of treatment at 3, 6 and 12 months
  Pulmonary function tests was performed, including the forced expiratory volume in 1 second (FEV1), to evaluated ventilation function at baseline and the end of treatment at 3, 6 and 12 Months.
Change from Baseline in the forced expiratory volume in 1 second of predicted (FEV1%pred) at 3, 6 and 12 Months. | From enrollment to the end of treatment at 3, 6 and 12 months
  Pulmonary function tests was performed, including the forced expiratory volume in 1 second of predicted (FEV1%pred), to evaluated ventilation function at baseline and the end of treatment at 3, 6 and 12 Months.
Change from Baseline in the FEV1/FVC ratio at 3, 6 and 12 Months. | From enrollment to the end of treatment at 3, 6 and 12 months
  Pulmonary function tests was performed, including the FEV1/FVC ratio, to evaluated ventilation function at baseline and the end of treatment at 3, 6 and 12 Months.
Change of the BNP/NT-Pro BNP from baseline to the end of treatment at 3, 6 and 12 months. | From enrollment to the end of treatment at 3, 6 and 12 months.
  The BNP/NT-Pro BNP will be measured at baseline the end of treatment at 3, 6 and 12 months to evaluate the condition of heart failure.
The restenosis rate of blood vessels after interventional therapy at the end of treatment at 3 and 12 months | From enrollment to the end of treatment at 3 and 12 months.
  Restenosis following interventional therapy was monitored at the end of treatment at 3 and 12 months, with restenosis defined as a blood vessel diameter reduction of more than 50% from the original size, or when the pressure gradient (Pd) at the site of vascular stenosis increases by 5 mmHg or more compared to the last measurement.
Change of the mediastinal lesion volume from baseline to 3 and 12 months after the end of treatment. | From enrollment to the end of treatment at 3 and12 months.
  The mediastinal lesion volume will be measured at baseline and 3, 12 months after the end of treatment using CTPA or PET-CT imaging. The volume is represented by the maximum transverse diameter of the cross-section of the lesion site.
Change from baseline of the quality-of-life score at 3, 6 and 12 months after the end of treatment. | From enrollment to the end of treatment at 3, 6 and 12 months
  Quality of life was assessed using the 36-Item Short-Form Health Survey (SF-36) at baseline and 3, 6 and 12 months after the end of treatment. The SF-36 scoring scale consists of 8 dimensions, which can be summarized as physical health and mental health. The score range of each dimension is 0 to 100 points. The higher the score, the better the health condition.
Number of participants with complications of bronchoscopy and pulmonary intervention. | Immediately or in the short term after treatment, and within 12 months after treatment
  Measure the probability of complications occurring during or after therapeutic operations. Complications of pulmonary vascular intervention include pulmonary vascular injury, arrhythmia, reperfusion pulmonary edema, etc; Complications of bronchoscopy include pneumothorax, massive hemoptysis, infection, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia M, Su H, Jiang K, Wang A, Guo Z, Zhu H, Zhang F, Sun X, Shi Y, Pan X, Cao Y. Incidence and predictors of in-stent restenosis following intervention for pulmonary vein stenosis due to fibrosing mediastinitis. Orphanet J Rare Dis. 2024 Oct 14;19(1):379. doi: 10.1186/s13023-024-03391-8. PMID 39397011
- [Background] Varghese C, Johnson GB, Eiken PW, Edell ES, Specks U, Larson NB, Peikert T. A Retrospective Evaluation of the Treatment Effects of Rituximab in Patients with Progressive and Symptomatic Fibrosing Mediastinitis. Ann Am Thorac Soc. 2024 Nov;21(11):1533-1541. doi: 10.1513/AnnalsATS.202405-533OC. PMID 39106522